CLINICAL TRIAL: NCT03918590
Title: Pain Control Following Intravitreal Injection Using Topical Nepefanac 0.3% or Pressure Patching: A Prospective, Randomized, Placebo Controlled Trial
Brief Title: Post Intravitreal Injection Topical NSAID vs. Patching
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The New York Eye & Ear Infirmary (Other)
Responsible Party: Principal Investigator, Ronald Gentile, MD, Professor, The New York Eye & Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16.15
Record Dates: First submitted 2019-04-04; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Neovascular Age-related Macular Degeneration; Diabetic Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — nepafenac; Suspensions; methylacetylene

STUDY DESIGN:
Intervention Model Description: Group 1: Placebo (Preservative free artificial tears) Group 2: Nepefanac 0.3% suspension Group 3: Patch for 2 hours
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- A single drop of nepafenac 0.3% suspension (Active Comparator): A single drop of nepafenac 0.3% suspension (Ilevro; Alcon, Fort Worth, TX)
  Interventions: Drug: nepafenac 0.3% suspension (Ilevro; Alcon, Fort Worth, TX)
- Patching (Other): A light pressure patch applied for two hours
  Interventions: Other: patching
- A single drop of preservative-free Artificial Tears (Placebo Comparator): A single drop of preservative-free Theratears tear drop, (Akron, Ann Arbor, MI).
  Interventions: Drug: Theratears tear drop, (Akron, Ann 111 Arbor, MI)

INTERVENTIONS:
Drug: nepafenac 0.3% suspension (Ilevro; Alcon, Fort Worth, TX) — NSAID
  Arms: A single drop of nepafenac 0.3% suspension
Drug: Theratears tear drop, (Akron, Ann 111 Arbor, MI) — preservative-free Artificial Tears
  Arms: A single drop of preservative-free Artificial Tears
Other: patching — no drug/ patching
  Arms: Patching

SUMMARY:
A prospective randomized trial, to evaluate post-injection comfort measures comparing topical NSAID (nepafenac 0.3% suspension) and patching.

DETAILED DESCRIPTION:
This is a single masked, randomized, placebo-controlled study that will enroll approximately 60 subjects with recent active retina related disease requiring intravitreal agents. Subjects will be randomized into one of 3 groups in a 1:1:1 ratio, and assigned to receive nepafenac 0.3% suspension or a sham procedure. Subjects will have a one in three (33%) chance of receiving active treatment (no sham procedure), a one in three (33%) chance of receiving patching procedure (no active treatment) or a one in three (33%) chance of receiving placebo (no active treatment).

Study participants will then complete the Visual Analog Scale immediately following injection and then after 1 hour, and, 24 hours. The VAS data along with relevant data related to each subject's injection will also be compiled, including, but not limited to: drug injected, diagnosis, co-morbid conditions, history of previous injections, visual acuity, age, and gender.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Already scheduled for anti-VEGF injection based on standard of care for disease process.
* Ability to provide written informed consent
* Capable of complying with study protocol.
* Volunteer written informed consent with the understanding that consent may be withdrawn by the subject at any time without prejudice to future care

Exclusion Criteria:

* History of past intraocular injection of steroid medication.
* Experiencing baseline eye pain
* Monocular; non-study eye with VA<20/100.
* Unwilling or unable to follow or comply with all study related procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-06-03 (Estimated)

PRIMARY OUTCOMES:
Post Intravitreal Injection Measurement of Pain | 6 hours and 24 hours after intravitreal injection
  Change from Baseline post intravitreal injection pain at 6 and 24 hours as measured by the Numeric Pain Rating Scale. The pain numeric rating scale (NRS), on which patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain"), at the screening, 6 hours and 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- New York Eye and Ear Infirmary, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No